CLINICAL TRIAL: NCT05857280
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Patients With Multiple Sclerosis (EXOSEP 2)
Brief Title: EXOPULSE Mollii Suit, Motor Function & Multiple Sclerosis (EXOSEP 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Shakhbout Medical City (Other)
Responsible Party: Principal Investigator, Naji Joseph Riachi, Principal Investigator, Sheikh Shakhbout Medical City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EXOSEP2
Record Dates: First submitted 2023-03-30; First posted 2023-05-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Sclerosis, Multiple; MS (Multiple Sclerosis); Spasticity, Muscle; Spastic
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXOPULSE Mollii Suit Stimulation Active (Active Comparator): This will be the EXOPULSE Mollii Suit Active Stimulation. Stimulation will go on for 60 minutes while control unit is on for 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation
- EXOPULSE Mollii Suit Stimulation Sham (Sham Comparator): This will be the EXOPULSE Mollii Suit Sham Stimulation. Stimulation will go on for 1 minute then it turns off while the control unit will remain on for total of 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation

INTERVENTIONS:
Device: EXOPULSE Mollii Suit Stimulation — We designed a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of motor functions and MS related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit stimulation. in phase 1, the patient will receive two stimulations separated by a two-week washout period. The patients will be randomized to receive either active/sham or sham/active and both patients and investigators will be blinded to the order in which the stimulation will be given. A 2-week washout period should be enough to prevent a potential carry over effect. Two weeks after the end of phase 1, a second open label phase (phase 2) of this trial will be proposed to all patients where they will receive active stimulation every other day at home over four weeks (for a total of 14 sessions). This will help understand the long term effects of EXOPULSE Mollii suit stimulation on MS related symptoms.

SUMMARY:
The goal of this clinical trial is to demonstrate the improvement of motor functions related symptoms in patients with MS and spasticity using Exopulse Mollii suit stimulation in Multiple Sclerosis patients with spasticity. The main questions it aims to answer are:

* to evaluate the short-term impact of EXOPULSE Mollii suit on balance in adult MS patients suffering from spasticity.
* to assess the effects of EXOPULSE Mollii suit on mobility, upper and lower limbs muscle tone, pain, fatigue and quality of life.

Participants will participate in:

* One baseline visit for inclusion during which the patient will undergo the first session (active or sham) along with evaluations (before and after the session)
* One visit after two weeks during which the patient will undergo the second session (active or sham) along with evaluations (before and after the session)
* One visit after two weeks of the second stimulation condition; the patients will undergo a third evaluation and receive the EXOPULSE Mollii Suit for the four-week open label phase and will use the suit at home for an active stimulation session every other day for four weeks.
* One visit at the end of the open label phase to perform the fourth and last evaluation and return the EXOPULSE Mollii suit.

Researchers will compare both Active and Sham groups to demonstrate the improvement of motor functions related symptoms in patients with MS and spasticity using Exopulse Mollii suit.

DETAILED DESCRIPTION:
The study is a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of motor functions and MS related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit stimulation. in phase 1, the patient will receive two stimulations separated by a two-week washout period. The patients will be randomized to receive either active/sham or sham/active and both patients and investigators will be blinded to the order in which the stimulation will be given. A 2-week washout period should be enough to prevent a potential carry over effect. Two weeks after the end of phase 1, a second open label phase (phase 2) of this trial will be proposed to all patients where they will receive active stimulation every other day at home over four weeks (for a total of 14 sessions). This will help understand the long term effects of EXOPULSE Mollii suit stimulation on MS related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis according to the 2017 McDonald criteria since at least one month.
* Age between 18 and 75 years.
* Ability to walk freely or with the need of support (expanded disability status scale score (EDSS) < 7).
* Being free of relapses in the last three months.
* Being able to understand verbal instructions.
* Having spasticity with a score of at least 1+ on the MAS.
* Having a BBS score ≤46 associated in the literature with a risk of fall.

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitor for the study purposes due to geographical or social reasons.
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump or other contraindications to using EXOPULSE Mollii suit.
* Being pregnant.
* Having a change in their pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 kg/m^2.
* In case of the introduction of a medical device other than EXOPULSE Mollii suit during the study period.
* Patients under juridical protection.
* Prisoners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Balance using Berg Balance Scale (BBS) | To be assessed at baseline.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in Patients with Multiple Sclerosis (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 2.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in Patients with Multiple Sclerosis (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 4.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in Patients with Multiple Sclerosis (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 8.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in Patients with Multiple Sclerosis (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.

SECONDARY OUTCOMES:
Visual Analog Score for spasticity. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Spasticity will be measured using a visual analog score from 0 to 10, 0 being no spasticity and 10 being the worst possible spasticity.
Mobility. | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
  Mobility will be evaluated by the 12-item Multiple Sclerosis Walking Scale (MSWS-12). Each one of the 12 items will be assessed and assigned numbers from 1 to 5, 1 being not at all to 5 being extremely common, and the results will be added to a total of 60, so the higher the score, the better the mobility.
Visual Analog Score for pain. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Pain will be measured using a visual analog score from 0 to 10, 0 being no pain, to 10 being the worst possible pain.
Multiple Sclerosis International Quality of Life Questionnaire. | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
  Quality of life will be measured using the 31-item Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL). This questionnaire consists of 31 questions covering 9 domains including: 1- activity of daily living; 2- physical well-being; 3- relationships with friends; 4- symptoms; 5- relationships with family; 6- relationships with health care systems; 7- sentimental and sexual life; 8- coping; and 9- rejection. The questions are answered by ticking or checking the box that describes best of what patients would feel ranging from 0 to 4, 0 being not at all and 4 always or very much.
  For MusiQoL, the score of each of the nine sub domains is calculated as the average for the set of questions making up the domain. An overall score is then calculated as the average of all the scores for each subdomain. Prior to computing the final overall score, each domain-specific score is linearly transformed to a 0-100 scale with 0 being the worst quality of life and 100 the best.
Overall Clinical improvement. | This to be assessed at baseline, then at week 2, and week 8.
  Evaluation of overall Clinical improvement will be done using the 7-point Clinical Global Impression (CGI). Patient will fill a questionnaire that will address their clinical situation as follows:
  1. Very much improved.
  2. Much improved.
  3. Slightly improved.
  4. No change.
  5. Slightly worse.
  6. Much worse.
  7. Very much worse.
  The score will range from 1-7, 1 being the best clinical outcome and 7 the worst.
Blinding Questionnaire. | This to be assessed at baseline, then at week 2.
  Evaluation of patient's blinding to the type of stimulation in the crossover trial periods using a dedicated questionnaire. Patients will be asked whether they think they received the sham or active stimulation.
  No scale will be used for this measure.
Visual Analog Score for fatigue. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Fatigue will be measured using a visual analog score from 0 to 10, 0 being no fatigue, to 10 being the worst possible fatigue.
Muscle tone. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Muscle tone will be evaluated by the Modified Ashworth Scale (MAS). Scores will range from 0 to 4, 0 being no increase or normal muscle tone, to 4 being rigidity in flexion or extension of muscles.
Fall Risk | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
  Fall risk will be assessed using the Falls Efficacy Scale-International scale. It is a 16-item scale, including a range of functional activities, that assesses the perceived risk of falling, using a score that will range from 1 to 4, 1 being not at all concerned to 4 being very concerned.
  Items are summed to a total score that will range from a minimum of 16 (no concern about falling) to a maximum of 64 (severe concern about falling).
Weight. | Baseline
  The patient weight will be measured and recorded in kilograms.
Height. | Baseline
  The patient height will be measured and recorded in centimeters.
Time Up and Go (TUG) | Baseline, and through study completion
  Patients have to stand up from a chair when they hear the verbal instruction "go", walk a distance of 3 meters, turn around, walk back to the chair and sit down. Timing starts with the verbal instruction "go' and stops when the patients return to the seated position. The score consists of the time taken to complete the test activity, measured in seconds.
Body Mass Index (BMI) | Baseline
  The weight and height will be combined to report BMI in kg/m^2. BMI of 35 kg/m^2 or more will be used as an exclusion criterion for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- SSMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andringa A, van de Port I, van Wegen E, Ket J, Meskers C, Kwakkel G. Effectiveness of Botulinum Toxin Treatment for Upper Limb Spasticity Poststroke Over Different ICF Domains: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2019 Sep;100(9):1703-1725. doi: 10.1016/j.apmr.2019.01.016. Epub 2019 Feb 21. PMID 30796921
- [Background] Arroyo R, Massana M, Vila C. Correlation between spasticity and quality of life in patients with multiple sclerosis: the CANDLE study. Int J Neurosci. 2013 Dec;123(12):850-8. doi: 10.3109/00207454.2013.812084. Epub 2013 Jul 15. PMID 23819835
- [Background] Bakaniene I, Urbonaviciene G, Janaviciute K, Prasauskiene A. Effects of the Inerventions method on gross motor function in children with spastic cerebral palsy. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):581-586. doi: 10.1016/j.pjnns.2018.07.003. Epub 2018 Jul 20. PMID 30061001
- [Background] Bar-On L, Molenaers G, Aertbelien E, Van Campenhout A, Feys H, Nuttin B, Desloovere K. Spasticity and its contribution to hypertonia in cerebral palsy. Biomed Res Int. 2015;2015:317047. doi: 10.1155/2015/317047. Epub 2015 Jan 11. PMID 25649546
- [Background] Baude M, Nielsen JB, Gracies JM. The neurophysiology of deforming spastic paresis: A revised taxonomy. Ann Phys Rehabil Med. 2019 Nov;62(6):426-430. doi: 10.1016/j.rehab.2018.10.004. Epub 2018 Nov 28. PMID 30500361
- [Background] Beard S, Hunn A, Wight J. Treatments for spasticity and pain in multiple sclerosis: a systematic review. Health Technol Assess. 2003;7(40):iii, ix-x, 1-111. doi: 10.3310/hta7400. PMID 14636486
- [Background] Bennett SE, Bromley LE, Fisher NM, Tomita MR, Niewczyk P. Validity and Reliability of Four Clinical Gait Measures in Patients with Multiple Sclerosis. Int J MS Care. 2017 Sep-Oct;19(5):247-252. doi: 10.7224/1537-2073.2015-006. PMID 29070965
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Burke D, Wissel J, Donnan GA. Pathophysiology of spasticity in stroke. Neurology. 2013 Jan 15;80(3 Suppl 2):S20-6. doi: 10.1212/WNL.0b013e31827624a7. PMID 23319482
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Christine C, Dolk H, Platt MJ, Colver A, Prasauskiene A, Krageloh-Mann I; SCPE Collaborative Group. Recommendations from the SCPE collaborative group for defining and classifying cerebral palsy. Dev Med Child Neurol Suppl. 2007 Feb;109:35-8. doi: 10.1111/j.1469-8749.2007.tb12626.x. No abstract available. PMID 17370480
- [Background] Cattaneo D, Regola A, Meotti M. Validity of six balance disorders scales in persons with multiple sclerosis. Disabil Rehabil. 2006 Jun 30;28(12):789-95. doi: 10.1080/09638280500404289. PMID 16754576
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] Ertzgaard P, Alwin J, Sorbo A, Lindgren M, Sandsjo L. Evaluation of a self-administered transcutaneous electrical stimulation concept for the treatment of spasticity: a randomized placebo-controlled trial. Eur J Phys Rehabil Med. 2018 Aug;54(4):507-517. doi: 10.23736/S1973-9087.17.04791-8. Epub 2017 Oct 25. PMID 29072043
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fernandez O, Costa-Frossard L, Martinez-Gines M, Montero P, Prieto JM, Ramio L. The Broad Concept of "Spasticity-Plus Syndrome" in Multiple Sclerosis: A Possible New Concept in the Management of Multiple Sclerosis Symptoms. Front Neurol. 2020 Mar 17;11:152. doi: 10.3389/fneur.2020.00152. eCollection 2020. PMID 32256440
- [Background] Flachenecker P, Henze T, Zettl UK. Spasticity in patients with multiple sclerosis--clinical characteristics, treatment and quality of life. Acta Neurol Scand. 2014 Mar;129(3):154-62. doi: 10.1111/ane.12202. Epub 2013 Nov 20. PMID 24256407
- [Background] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Background] Goldenberg MM. Multiple sclerosis review. P T. 2012 Mar;37(3):175-84. No abstract available. PMID 22605909
- [Background] Gupta AD, Chu WH, Howell S, Chakraborty S, Koblar S, Visvanathan R, Cameron I, Wilson D. A systematic review: efficacy of botulinum toxin in walking and quality of life in post-stroke lower limb spasticity. Syst Rev. 2018 Jan 5;7(1):1. doi: 10.1186/s13643-017-0670-9. PMID 29304876
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Henze T, Rieckmann P, Toyka KV; Multiple Sclerosis Therapy Consensus Group of the German Multiple Sclerosis Society. Symptomatic treatment of multiple sclerosis. Multiple Sclerosis Therapy Consensus Group (MSTCG) of the German Multiple Sclerosis Society. Eur Neurol. 2006;56(2):78-105. doi: 10.1159/000095699. Epub 2006 Sep 8. PMID 16966832
- [Background] Hughes C, Howard IM. Spasticity management in multiple sclerosis. Phys Med Rehabil Clin N Am. 2013 Nov;24(4):593-604. doi: 10.1016/j.pmr.2013.07.003. PMID 24314678
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Mai J, Pedersen E. Mode of action of dantrolene sodium in spasticity. Acta Neurol Scand. 1979 Jun;59(6):309-16. doi: 10.1111/j.1600-0404.1979.tb02941.x. PMID 158280
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Background] Mukherjee A, Chakravarty A. Spasticity mechanisms - for the clinician. Front Neurol. 2010 Dec 17;1:149. doi: 10.3389/fneur.2010.00149. eCollection 2010. PMID 21206767
- [Background] Nielsen JB, Petersen NT, Crone C, Sinkjaer T. Stretch reflex regulation in healthy subjects and patients with spasticity. Neuromodulation. 2005 Jan;8(1):49-57. doi: 10.1111/j.1094-7159.2005.05220.x. PMID 22151383
- [Background] Nordstrom B, Prellwitz M. A pilot study of children and parents experiences of the use of a new assistive device, the electro suit Mollii. Assist Technol. 2021 Sep 3;33(5):238-245. doi: 10.1080/10400435.2019.1579267. Epub 2019 Apr 4. PMID 30945989
- [Background] Palmcrantz S, Pennati GV, Bergling H, Borg J. Feasibility and potential effects of using the electro-dress Mollii on spasticity and functioning in chronic stroke. J Neuroeng Rehabil. 2020 Aug 10;17(1):109. doi: 10.1186/s12984-020-00740-z. PMID 32778118
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Perrot A, Castanier C, Maillot P, Zitari H. French validation of the modified-falls efficacy scale (M-FES Fr). Arch Gerontol Geriatr. 2018 Sep-Oct;78:233-239. doi: 10.1016/j.archger.2018.07.001. Epub 2018 Jul 4. PMID 30025268
- [Background] Picelli A, Santamato A, Chemello E, Cinone N, Cisari C, Gandolfi M, Ranieri M, Smania N, Baricich A. Adjuvant treatments associated with botulinum toxin injection for managing spasticity: An overview of the literature. Ann Phys Rehabil Med. 2019 Jul;62(4):291-296. doi: 10.1016/j.rehab.2018.08.004. Epub 2018 Sep 13. PMID 30219307
- [Background] Pozzilli C. Overview of MS spasticity. Eur Neurol. 2014;71 Suppl 1:1-3. doi: 10.1159/000357739. Epub 2014 Jan 22. No abstract available. PMID 24457845
- [Background] Pugliatti M, Rosati G, Carton H, Riise T, Drulovic J, Vecsei L, Milanov I. The epidemiology of multiple sclerosis in Europe. Eur J Neurol. 2006 Jul;13(7):700-22. doi: 10.1111/j.1468-1331.2006.01342.x. PMID 16834700
- [Background] Rabchevsky AG, Kitzman PH. Latest approaches for the treatment of spasticity and autonomic dysreflexia in chronic spinal cord injury. Neurotherapeutics. 2011 Apr;8(2):274-82. doi: 10.1007/s13311-011-0025-5. PMID 21384222
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Sidovar MF, Limone BL, Coleman CI. Mapping of Multiple Sclerosis Walking Scale (MSWS-12) to five-dimension EuroQol (EQ-5D) health outcomes: an independent validation in a randomized control cohort. Patient Relat Outcome Meas. 2016 Feb 3;7:13-8. doi: 10.2147/PROM.S96956. eCollection 2016. PMID 26893584
- [Background] Stevenson T. Berg balance test. Phys Ther. 1996 Oct;76(10):1124, 1126. doi: 10.1093/ptj/76.10.1124. No abstract available. PMID 8863765
- [Background] Toomey E, Coote S. Between-rater reliability of the 6-minute walk test, berg balance scale, and handheld dynamometry in people with multiple sclerosis. Int J MS Care. 2013 Spring;15(1):1-6. doi: 10.7224/1537-2073.2011-036. PMID 24453756
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Rammohan KW, Rosenberg JH, Lynn DJ, Blumenfeld AM, Pollak CP, Nagaraja HN. Efficacy and safety of modafinil (Provigil) for the treatment of fatigue in multiple sclerosis: a two centre phase 2 study. J Neurol Neurosurg Psychiatry. 2002 Feb;72(2):179-83. doi: 10.1136/jnnp.72.2.179. PMID 11796766
- [Background] van Vliet R, Hoang P, Lord S, Gandevia S, Delbaere K. Falls efficacy scale-international: a cross-sectional validation in people with multiple sclerosis. Arch Phys Med Rehabil. 2013 May;94(5):883-9. doi: 10.1016/j.apmr.2012.10.034. Epub 2012 Dec 13. PMID 23246897
- [Background] Vivancos-Matellano F, Pascual-Pascual SI, Nardi-Vilardaga J, Miquel-Rodriguez F, de Miguel-Leon I, Martinez-Garre MC, Martinez-Caballero I, Lanzas-Melendo G, Garreta-Figuera R, Garcia-Ruiz PJ, Garcia-Bach M, Garcia-Aymerich V, Bori-Fortuny I, Aguilar-Barbera M; Spanish Group on Spasticity. [Guide to the comprehensive treatment of spasticity]. Rev Neurol. 2007 Sep 16-30;45(6):365-75. Spanish. PMID 17899519